CLINICAL TRIAL: NCT05556837
Title: Effect of Extruded Cereals Enriched With β-glucan From Oats or Barley on Postprandial Plasma Glucose and Serum Insulin Responses in Generally Healthy Adults
Brief Title: Effect of Extruded Cereals Enriched With β-glucan on Postprandial Plasma Glucose and Serum Insulin Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: INQUIS Clinical Research (Industry); Cereal Partners Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: INQ-2203
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Postprandial glucose; Postprandial insulin; Beta Glucan; Oats; Barley

STUDY DESIGN:
Intervention Model Description: The study is a double-blinded, randomized, crossover design with all subjects completing all 3 tests.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be double-blinded; the participants, those serving the participants and those doing the biochemical analysis, entering data, and performing the statistical analysis will be blinded to the nature of the test meals.
  The codes identifying the test meals will be kept in a sealed opaque envelope at INQUIS and will be opened only if necessary to assist in the diagnosis and management of a serious adverse event. Test meal identity on study documents and blood tubes will be the code numbers on the test food packages. Thus, the identity of the test meals will be double-blinded. The codes will be broken once the database for plasma glucose and serum insulin has been cleaned, locked, and sent to the sponsor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Cereal (Placebo Comparator): A portion of cereal (25g available carbohydrate) that contains no beta-glucan
  Interventions: Other: Control Cereal
- OBG Cereal (Experimental): A portion of cereal (25g available carbohydrate) that contains approximately 1.4g of oat beta-glucan (OBG)
  Interventions: Other: OBG Cereal
- BBG Cereal (Experimental): A portion of cereal (25g available carbohydrate) that contains approximately 1.4g of barley beta-glucan (BBG)
  Interventions: Other: BBG Cereal

INTERVENTIONS:
Other: Control Cereal — A portion of cereal (25g available carbohydrate), served with 125ml of 2% milk and 250ml water, will be fed to participants and postprandial glucose and insulin will be measured
  Arms: Control Cereal
Other: OBG Cereal — A portion of cereal (25g available carbohydrate) containing OBG, served with 125ml of 2% milk and 250ml of water, will be fed to participants and postprandial glucose and insulin will be measured
  Arms: OBG Cereal
Other: BBG Cereal — A portion of cereal (25g available carbohydrate) containing BBG, served with 125ml of 2% milk and 250ml of water, will be fed to participants and postprandial glucose and insulin will be measured
  Arms: BBG Cereal

SUMMARY:
β-glucan (BG) is a viscous dietary fiber present in barley and oats that, when added to carbohydrate containing foods, reduces the postprandial glycemic response (PPGR), which is considered to be beneficial to health. In 2011, the European Food Safety Authority (EFSA) concluded that 4g of either oat BG (OBG) or barley BG (BBG) per 30g available carbohydrate (avCHO) is required to obtain a reduction in PPGR, however this is an impractically large amount of BG to incorporate into palatable foods. A recent systematic review and meta-analysis found that doses of OBG well below 4g/30g avCHO can significantly reduce PPGR.

It is therefore hypothesized that 25g avCHO portions of cereal containing 1.4-1.5g of either OBG or BBG will elicit a statistically significantly lower PPGR compared to a control cereal containing no BG.

DETAILED DESCRIPTION:
Statistical Analysis:

Analysis populations: The intention-to-treat (ITT) population includes all subjects who consumed at least 1 of the 3 test meals in that phase. The per-protocol (PP) population for each phase includes all subjects who completed all 3 tests in that phase with no serious protocol violations. There may also be a group, termed PPDO (dropouts), defined as the PP population plus subjects who competed 1 or 2 of the 3 tests with no serious protocol violations.

Conclusions will be based on the glucose and insulin endpoints for the PP population. To assess the potential impact of excluding those subjects who dropped out after completing 1 or 2 tests, a secondary analysis will be performed for the PP+DO population where the missing values are imputed using methods described by Snedecor and Cochran.

Distribution of data: the methods of analyzing continuous data assume that the data are normally distributed. Normality of distribution will be tested by comparing the actual distribution of the Z scores to the expected distribution using the chi-square test with the data taken to be normally distributed if p>0.05. Non-normally distributed data will be transformed by (in order of preference) log-transformation, square-root-transformation, some other method, until the transformed data are normally distributed.

Primary endpoint: the primary endpoint will be assessed as follows: serum glucose concentrations will be subjected to repeated-measures analysis of variance (ANOVA) using the linear model analyzing for the main effects of time and treatment and the time×treatment interaction. After demonstrating a significant time×treatment interaction (indicating that the pattern of glucose response differs significantly among treatments), the values for iAUC 0-2h will be analyzed by ANOVA for the main effect of treatment; after demonstrating significant heterogeneity, the mean for each of the 2 test cereals will be compared only to that of each respective control cereal using Dunnett's Test to adjust for multiple comparisons. The 2 test cereals will not be compared to each other. The criterion for significance will be two-tailed p<0.05.

Secondary endpoints: the results for insulin iAUC will be assessed as described for the primary endpoint. Serum glucose and insulin concentrations and increments at each time point will be subjected to repeated-measures ANOVA. Upon demonstration of significant heterogeneity, individual means of the test and matched control cereals will be compared using Dunnett's Test to adjust for multiple comparisons. The 2 test cereals will not be compared to each other. The criterion for significance will be two-tailed p<0.05.

Statistical Power:

The average within-individual CV of glucose iAUC elicited by repeated tests of oral glucose is within the range of 22-25% in our previous studies in healthy individuals. To demonstrate that both test cereals differ significantly from the control, each comparison must have 90% power to detect a significant difference in order to obtain 80% power to detect both significant differences (since 0.902 = 0.81). Assuming a SD of 25% and using the normal distribution, n=40 subjects provide 95% power to detect a significant difference of 20% between test and control cereals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are non-pregnant, non-lactating aged 20-65 years of age, inclusive.
* Body mass index 18.0 to 29.9 kg/m², inclusive.
* Nonsmokers (tobacco, cannabis, vaping).
* Fasting glucose concentration <7.0 mmol/L (126 mg/dL), determined by a fasting finger-stick blood sample (plasma) at screening.
* Willing to abstain from unusual levels of food intake, unusual or strenuous exercise, smoking or consuming alcoholic drinks 24 hours before study days.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.
* Willing to comply with the protocol.
* Subjects must be eligible to receive income in Canada and be covered by a health insurance plan such as the Ontario Health Insurance Plan.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria.
* Systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg at screening.
* Change in body weight of >3.5kg (>7.7 lbs.) within 4 weeks of the screening visit.
* Practicing any extreme dietary habits, as judged by the Investigator (i.e., Atkins diet, very high protein diet, etc.).
* Major trauma or major medical or surgical event within 3 months of screening.
* History or presence of clinically important endocrine, cardiovascular, pulmonary, biliary, or gastrointestinal disorders.
* The use of medications known to influence carbohydrate metabolism, including, but not limited to adrenergic blockers, thiazolidinediones, metformin, and systemic corticosteroids, or with any condition or use of any medication which might, in the opinion of the Qualified Investigator (QI), either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Use of supplements containing chromium (intended for glucose management), ginseng or cinnamon, within 3 weeks of screening.
* Changes in the doses of permissible prescription drugs within 3 months of screening or changes in the doses of over-the-counter drugs or permissible supplements within 3 weeks of screening.
* History of cancer in the prior two years, except for non-melanoma skin cancer.
* Recent history (within 12 months of screening) or strong potential for alcohol or substance abuse, where alcohol abuse is defined as > 14 drinks per week (1 drink=12 oz beer, 5 oz wine, or 1.5 oz distilled spirits).
* Known intolerance, sensitivity, or allergy to any ingredients in the study test meals.
* Unwillingness or inability to comply with the experimental procedures and to follow INQUIS health and safety policies.
* Subject is currently participating or recently (within 30 days of screening) participated in a clinical trial involving long-term exposure (greater than 24 hours) to an investigational drug, nutritional supplement, or lifestyle modification.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Postprandial Glucose Incremental Area under the Curve (iAUC) from 0-2 hours | Plasma glucose will be measured for 2 hours after consumption of the cereals (timepoints: -5, 0, 15, 30, 45, 60, 90, and 120 minutes)
  iAUC, ignoring area below baseline, will be calculated from glucose concentrations in plasma obtained from finger prick blood samples. The mean glucose concentration at -5 and 0 minutes will be taken as the baseline.

SECONDARY OUTCOMES:
Postprandial Insulin iAUC from 0-2 hours | Serum insulin will be measured for 2 hours after consumption of the cereals (timepoints: -5, 0, 15, 30, 45, 60, 90, and 120 minutes)
  iAUC, ignoring area below baseline, will be calculated from insulin concentrations in serum obtained from finger prick blood samples. The mean insulin concentration at -5 and 0 minutes will be taken as the baseline.
Peak Rise of glucose | Glucose will be measured over 2 hours postprandially (timepoints: -5, 0, 15, 30, 45, 60, 90, and 120 minutes)
  the maximum postprandial increments (peak rises) of glucose defined as the maximum concentration achieved minus the baseline (mean of concentrations at -5 and 0 min)
Peak Rise of insulin | Insulin will be measured over 2 hours postprandially (timepoints: -5, 0, 15, 30, 45, 60, 90, and 120 minutes)
  the maximum postprandial increments (peak rises) of insulin defined as the maximum concentration achieved minus the baseline (mean of concentrations at -5 and 0 min)
Gmax | Glucose will be measured over 2 hours postprandially (timepoints: -5, 0, 15, 30, 45, 60, 90, and 120 minutes)
  The maximum postprandial concentration of glucose (Gmax) achieved over the 2h test period
Imax | Insulin will be measured over 2 hours postprandially (timepoints: -5, 0, 15, 30, 45, 60, 90, and 120 minutes)
  The maximum postprandial concentration of insulin (Imax) achieved over the 2h test period
Time of Gmax | Insulin will be measured over 2 hours postprandially (timepoints: -5, 0, 15, 30, 45, 60, 90, and 120 minutes)
  The time when the maximum postprandial concentration of glucose (Gmax) occurred during 2h test period
Time of Imax | Insulin will be measured over 2 hours postprandially (timepoints: -5, 0, 15, 30, 45, 60, 90, and 120 minutes)
  The time when the maximum postprandial concentration of insulin (Imax) occurred during 2h test period
Glucose concentrations and increments at each time point | Glucose will be measured over 2 hours postprandially (timepoints: -5, 0, 15, 30, 45, 60, 90, and 120 minutes)
  Glucose concentrations and increments at each time point
Insulin concentrations and increments at each time point | Glucose and insulin will be measured over 2 hours postprandially (timepoints: -5, 0, 15, 30, 45, 60, 90, and 120 minutes)
  Insulin concentrations and increments at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, DM, PhD, Principal Investigator — INQUIS Clinical Research
Locations (1):
- INQUIS Clinical Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No